CLINICAL TRIAL: NCT02202538
Title: Indego® Exoskeleton; Assessing Mobility for Persons With Spinal Cord Injury (SCI).
Acronym: Indego
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Hannifin Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-IND01
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Spinal Cord Injury
Keywords: SCI; Indego; Walking
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indego (Experimental): Indego
  Interventions: Device: Indego

INTERVENTIONS:
Device: Indego — Indego

SUMMARY:
This study will evaluate the Indego® device for safety and effectiveness at allowing persons with SCI who are non-ambulatory or poorly ambulatory to stand up and walk under a variety of conditions.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Height 5'1" to 6'3" (Acceptable height may vary by a few inches depending on femur length).
* Hip width as measured in sitting no greater than 16.6" (42 cm) (acceptable hip width may vary depending on soft tissue).
* Femur length as measured in sitting must be between 14 inches (35.5cm) and 18.5 inches (47 cm)
* Weight 250lbs (113.4 kg) or less
* Present with Spinal Cord Injury and NLI C5 and lower, with ISNCSCI A, B, C or D who are non-ambulatory or poorly ambulatory.
* There are no restrictions on time since injury. However, each subject must have signed medical clearance/approval for full weight bearing and locomotor training.
* Determined to have sufficient bone health for walking with full weight bearing without undue risk for fracture. Meeting of this criterion is at the discretion of each subject's personal MD and must be approved by each site's Medical PI.
* Passive range of motion (PROM) at shoulders, trunk, upper extremities and lower extremities within functional limits for safe gait and use of appropriate assistive device/stability aid.
* Skin must be intact where it interfaces with robotic device
* Modified Ashworth Scale for spasticity score must be 3 or less.
* Blood pressure and heart rate within established guidelines for locomotor training:

  * At rest; Systolic 150 or less Diastolic 90 or less and Heart rate 105 or less
  * Exercise; Systolic 180 or less Diastolic 105 or less and Heart Rate 145 or less
* Tolerate being in an upright standing position (passive or active) without being lightheaded or having a headache.

Exclusion Criteria:

* Weight in excess of 250 lbs
* Heterotopic ossification that, in the opinion of the investigator, would place the subject at undue risk for fracture.
* Any subject deemed at increased risk for injury by Medical Personnel
* Lower extremity joint limitation that exceeds 10 degrees at their hips, knees or ankles.
* Light headedness or headache in standing position (active or passive)
* Moderate to Severe Traumatic (or Acquired) Brain Injury
* Inability to follow instructions
* Colostomy bag
* Women who are pregnant or attempting to become pregnant during the study intervention.
* Unable to obtain informed consent (either from the subject or from the subjects Legally Authorized Representative).
* Any disease, concomitant injury, or condition that interferes with the performance or interpretation of the protocol specified assessments
* Unlikely to be available for follow-up phone call.
* Any other issue which, in the opinion of the investigators, will make the subject unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Craig Hospital, Englewood, Colorado
  - Shepherd Center, Atlanta, Georgia
  - Rehabilitation Institue of Chicago, Chicago, Illinois
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - RUSK Rehabilitation Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at five sites in the United States
Groups:
- All Subjects: All subjects enrolled in the study used the Indego
Period: Overall Study
Arm/Group | All Subjects
Started | 53
Screen Failure | 2
Completed | 45
Not Completed | 8
Not completed — Withdrawal by Subject | 5
Not completed — Did not meet all inclusion criteria | 2
Not completed — Investigator Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 53
Level of Injury [Number; unit: participants]
  T3 | 3
  T4 | 9
  T5 | 6
  T6 | 5
  T7 | 3
  T8 | 6
  T9 | 1
  T10 | 7
  T11 | 5
  T12 | 5
  L1 | 2
  L2 | 1
ASIA Impairment Scale Score [Number; unit: participants] — A: motor and sensory complete injury B: motor complete and sensory incomplete injury C: motor and sensory incomplete injury; half or more than half of affected muscles are less than grade 3/5 D: motor and sensory incomplete injury; half or more than half of affected muscles are more than grade 3/5
  Reference: rehabmeasures.org
  participants
    A | 36
    B | 5
    C | 11
    D | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Able to Complete the 600 Meter Walk Test (600MWT)
Description: Measured time for an individual to complete walking 600 meters on a level surface with the Indego and stability aid at the end of the study, proposed to be representative of an individual's ability to ambulate in the community.
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Groups:
- All Enrolled Subjects Who Completed the Study: All subjects in the study used the Indego
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
percentage of participants | 95.6

2. Primary Outcome: Average Speed of 10 Meter Walk Test (10MWT) Mid Study Versus End of Study
Description: Measured time for an individual to complete walking 10 meters with the Indego and a stability aid midway through the study and at the end of the study.
Time Frame: 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
meters/second
  Average speed for 10MWT mid study | 0.31 (0.10)
  Average speed for 10MWT end of study | 0.37 (0.09)

3. Primary Outcome: Timed Up and Go (TUG) Test
Description: Measures the time required for an individual to stand from a seated position, walk three meters, turn, walk back three meters, turn and return to a seated position.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
seconds | 84.09 (20.41)

4. Primary Outcome: Average Time to Don/Doff Device
Description: Time needed for an individual to don or doff the device.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
minutes
  Average time to don device | 9.3 (4.5)
  Average time to doff device | 2.6 (1.4)

5. Primary Outcome: Percentage of Subjects That Could Don/Doff the Device Independently
Description: The percentage of participants that could don/doff the device independently at the end of the study, without the help of their Physical Therapist.
Time Frame: 8 weeks
Measure: Number; unit: percentage
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
percentage
  Subjects that could don device independently | 62.2
  Subjects that could doff device independently | 82.2

6. Secondary Outcome: Walking Index for Spinal Cord Injury (WISCI-II) Assessment
Description: Assesses physical assistance and devices required for persons to walk following paralysis resulting from a Spinal Cord Injury.
  0:unable
  1. parallel bars, braces, help of 2 persons,<10m
  2. parallel bars, braces, help of 2 persons,10m
  3. parallel bars, braces, help of 1 person,10m
  4. parallel bars, no braces, help of 1 person,10m
  5. parallel bars, braces, no help,10m
  6. walker, braces, help of 1 person,10m 7:2 crutches, braces, help of 1 person,10m
  8:walker, no braces, help of 1 person,10m 9:walker, braces, no help,10m 10:1 cane/crutch, braces, help of 1 person,10m 11:2 crutches, no braces, help of 1 person,10m 12:2 crutches, braces, no help,10m 13:walker, no braces/help,10m 14:1 cane/crutch, no braces, help of 1 person,10m 15:1 cane/crutch, braces, no help,10m 16:2 crutches, no braces/help,10m 17:no devices/braces, help of 1 person,10m 18: no devices, braces, no help,10m 19:1cane/crutch, no braces/help,10m 20:no devices/braces/help,10m
  Reference: rehabmeasures.org
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
units on a scale | 6.8 (1.5)

7. Secondary Outcome: Functional Independence Measure (FIM) Score for Walking Indoors
Description: FIM measures an individual's level of disability and indicates how much assistance is needed for that individual to carry out activities of daily living.
  7: complete independence 6: modified independence 5: supervision or setup assistance 4: minimal contact assistance 3: moderate assistance 2: maximal assistance
  1: total assistance
  Reference: rehabmeasures.org
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
units on a scale | 4.3 (0.5)

8. Secondary Outcome: Borg Rating of Perceived Exertion (BRPE) for Walking Indoors
Description: The BPRE characterizes the level of effort required by an individual to perform a task and takes into account both the person's fitness level and the difficulty of the task.
  6: no exertion at all 7: extremely light 8-9: very light 10-11: light 12-13: somewhat hard 14-15: hard (heavy) 16-17: very hard 18-19: extremely hard 20: maximal exertion
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Enrolled Subjects Who Completed the Study
Number analyzed (Participants) | 45
units on a scale | 10.4 (2.2)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 19/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=53)
Bruise (Skin and subcutaneous tissue disorders) | 6
Pain (Musculoskeletal and connective tissue disorders) | 3
Scrape/Cut/Abrasion (Skin and subcutaneous tissue disorders) | 10
Skin Redness (Skin and subcutaneous tissue disorders) | 3
Tachycardia (Cardiac disorders) | 4
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No